CLINICAL TRIAL: NCT03721692
Title: Remote Ischemic Conditioning in Acute Ischemic Cerebral Vascular Disease Patients With Coexistence of Cerebral and Coronary Atherosclerosis（RIC-CCCA）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigater, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIC-CCCA
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-03

CONDITIONS: Acute Ischemic Cerebral Vascular Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The patients will accept cardio-cerebrovascular disease secondary prevention treatment and use RIC everyday for three months, 5 cycles 5min ischemic-5min reperfusion each day.
  Interventions: Device: RIC
- non-RIC group (No Intervention): The patients will only accept cardio-cerebrovascular disease secondary prevention treatment.

INTERVENTIONS:
Device: RIC — The patients will use RIC everyday for three months, 5 cycles 5min ischemic-5min reperfusion each day.
  Arms: RIC group

SUMMARY:
Remote ischemic conditioning(RIC) is a protective systemic strategy by organs brief and sublethal ischemia to confer protection from subsequent severe ischemia in distant organs, especially for heart and brain. This study will discuss whether RIC can play a part in preventing the patients with coexistence of cerebral and coronary atherosclerosis from the recurrence of cerebral vascular disease(CVD) or coronary artery disease(CAD). This study selects patients who suffered an ischemic stroke within 14 days prior to enrollment. All patients complete cerebral and coronary artery assessment. And then the the investigators select the patients who both have at least one cerebral vascular and at least one coronary artery stenosis over 50%, or the patients who both have at least one cerebral vascular stenosis over 50% and myocardial ischemic events history. These patients will randomly divide into two groups, RIC group and non-RIC group. Non-RIC group will only accept cardio-cerebrovascular disease secondary prevention treatment. RIC group will use not only cardio-cerebrovascular disease secondary prevention treatment, but also RIC everyday for three months, 5 cycles 5min ischemic-5min reperfusion each day. For the first month, the the investigators will call RIC group patients every week for insuring compliance and adverse effect. All patients will follow up endpoint events, cardio-cerebrovascular disease secondary prevention treatment, and the adverse effect every three months, up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who suffered an ischemic stroke within 14 days prior to enrollment
2. With a baseline NIHSS score 0-15, mRS score 2-4
3. With at least one cerebral and carotid artery stenosis over 50%
4. With at least one coronary artery stenosis over 50% or previous myocardial ischemic events history(tertiary hospital doctors judge angina, myocardial infarction, and coronary revascularization treatment)
5. Age from 18 to 80
6. Informed consent obtained

Exclusion Criteria:

1. Thrombolytic therapy within 24 h prior to enrollment
2. Progressive neurological signs within 24 h prior to enrollment
3. Arterial stenosis due to unequivocal cardiac source of embolism, arterial dissection, vasculitic disease, cerebral venous thrombosis, Moyamoya disease
4. Arterial stenosis due to benign angiopathy of central nervous system, post-partum angiopathy, suspected vasospastic process, suspected recanalized embolus, neurosyphilis, any other intracranial infection
5. Rheumatic mitral disease with or without aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis
6. Uncontrolled severe hypertension, defined by sitting systolic blood pressure(SBP) > 180 mm Hg and/or sitting diastolic blood pressure(DBP) > 110 mm Hg after medication
7. Contraindication for remote ischemic conditioning, including severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs
8. Subclavian arterial stenosis 50% or subclavian steal syndrome
9. Severe hemostatic disorder or severe coagulation dysfunction, platelets < 100 ×10^9/L
10. Aspartate aminotransferase(AST) and/or Alanine aminotransferanse(ALT) > 3× the upper limit of the reference range; creatinine clearance < 0.6 mL/s and/or serum creatinine > 265 mmol/L (>3.0 mg/dL)
11. Unwilling to comply with the treatment or follow-up assessments
12. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, or epidural) within 90 days prior to enrollment
13. Intracranial neoplasm, cerebral aneurysm, or arteriovenous malformation
14. Retinal hemorrhage or visceral bleeding within 30 days prior to enrollment
15. Major surgery, including cardiac and open femoral, aortic, or carotid surgery, within 30 days prior to enrollment or intent to undergo within 12 months after enrollment
16. Life expectancy < 3 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Complex ischemic cardio-cerebrovascular events cumulative incidence | 1 year
  include non-fatal acute ischemic cerebral vascular disease, non-fatal acute coronary syndrome, cardio-cerebrovascular events lead to death, elective cardio-cerebralvascular revascularization, myocardial and cerebral ischemia lead to hospitalize

SECONDARY OUTCOMES:
Primary Outcome Events Occur | 1 year
  The first time of the primary outcome events occur
Rate of all-cause death | 1 year
  One year all-cause death rate
Score of Modified Rankin Scale(mRS) | 3 months
  The Modified Rankin Scale Score (mRS) is the most comprehensive and most widely used primary outcome measurement to assess the neurological functional disability in contemporary acute stroke trials. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranges from 0 (no symptom) to 5 (severe disability) and 6 (death). We will use mRS to evaluate the degree of disability or dependence during daily activities. The mRS will be assessed by certified study investigator at 3 months. The distribution of mRS will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China